CLINICAL TRIAL: NCT03059381
Title: Investigation of the Clinical Safety and Efficacy of Long-term Treatment With Fycompa Tablets in Adolescence Epilepsy Patients With Partial-onset Seizures (With or Without Secondary Generalized Seizures) or Primary Generalized Tonic-clonic Seizures
Acronym: FYC02T
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E2007-M081-503
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2021-04

CONDITIONS: Partial Seizures (With or Without Secondary Generalized Seizures); Primary Generalized Tonic-clonic Seizures
Keywords: adolescent epilepsy participants; partial seizures; primary generalized Tonic-clonic seizures
MeSH Terms: conditions — Seizures | interventions — perampanel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fycompa-treated epilepsy participants: Adolescent epilepsy participants with partial-onset seizures (with or without secondary generalized seizures) or primary generalized Tonic-clonic seizures who receive long-term treatment with Fycompa
  Interventions: Drug: Fycompa

INTERVENTIONS:
Drug: Fycompa — The usual oral dosage for adults and children 12 years of age or older is initially 2 milligrams (mg) once daily as perampanel at bedtime, and the daily dose may then be increased by 2 mg at intervals of 1 week or longer. The maintenance dose is 8 mg once daily in the absence of concomitant antiepileptic drugs that accelerate the metabolism of this product, or 8 to 12 mg once daily in the presence of such concomitant drugs. The dosage may be increased or decreased as necessary by 2 mg at intervals of 1 week or longer depending on symptoms, but the maximum daily dose should not be over 12 mg.

SUMMARY:
The objective of this study is to identify the following in adolescent epilepsy participants with partial-onset seizures (with or without secondary generalized seizures) or primary generalized Tonic-clonic seizures who receive long-term treatment with Fycompa:

1. unknown adverse drug reactions (ADRs);
2. occurrence of ADRs;
3. factors that are likely to affect safety and efficacy;
4. occurrence of dizziness, balance disorders, ataxia, muscle relaxation-related adverse events, and falls as priority investigation items;
5. occurrence of psychiatric adverse events as priority investigation items (eg, aggression).

ELIGIBILITY:
Inclusion Criteria:

* Epilepsy participants from 12 to 17 years of age with:

  * Partial seizures (with or without secondary generalized seizures)
  * Primary generalized Tonic-clonic seizures

Exclusion Criteria:

* Participants previously treated with Fycompa

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants with epilepsy who will receive Fycompa per the approved indication in routine clinical practice
Sampling Method: Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2021-03-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with any serious adverse event | from 0 to 104 weeks
Number of participants with any non-serious adverse event | from 0 to 104 weeks

SECONDARY OUTCOMES:
Number of participants experiencing seizures | from 0 to 104 weeks
Overall improvement rating in seizure frequency | from 0 to 104 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Inoue Y, Sumitomo K, Matsutani K, Ishii M. Real-world evaluation of perampanel effectiveness in Japanese adolescents with epilepsy. Epileptic Disord. 2022 Oct 1;24(5):813-821. doi: 10.1684/epd.2022.1454. PMID 35792849